CLINICAL TRIAL: NCT05358236
Title: The Effect of Episiotomy Wound Care and Genital Hygiene Training on Episiotomy Wound Healing and Pain Perception: Randomized Controlled Trial
Brief Title: Episiotomy Wound Care, Episiotomy Wound Healing and Pain Perception
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Gonca Buran, Principal Investigator, Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2022/4
Record Dates: First submitted 2022-04-26; First posted 2022-05-03 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2022-05

CONDITIONS: Episiotomy Wound; Wound Healing; Pain; Training, Toilet
Keywords: wound healing; Episiotomy; genital hygiene; postpartum care; REEDA scale
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: The research is an experimental study with parallel groups including randomized controlled, experimental, and control with educational intervention
Who Masked: Investigator, Outcomes Assessor
Masking Description: No intervention will be made by the responsible researcher. Thus, she will be blinded to the experimental and control groups. The training intervention and data collection process will be carried out by the co-researcher. It will also enter the data into the SPSS program as A and B groups. The analysis will be carried out by the researcher blinded to the groups. After the reporting process is completed, it will be announced to which groups A and B groups belong. Participants will also be blind to each other.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- training + written and illustrated training brochure (Other): Postpartum first day was given wound care and genital hygiene training (one hour).
  At the end of the training, the mothers were given a written and illustrated training brochure.
  Interventions: Other: Episiotomy Wound Care and Genital Hygiene Training
- Standard of care (Control group) (No Intervention): Standard of care (Control group) Left to the usual care of the hospital

INTERVENTIONS:
Other: Episiotomy Wound Care and Genital Hygiene Training — Episiotomy wound healing and genital hygiene training were given face-to-face by researchers to the mothers assigned to the training group. The trainings were given to each mother individually in their rooms. The total training lasted an average of one hour. At the end of the training, the mothers were given a written and illustrated training brochure.
  Training content
  * Primarily, external reproductive organs were shown to mothers through pictures.
  * Urethra, Vagina, Anus, Perineum areas were mentioned.
  * The definition of Episiotomy was made; and where and how it was applied was explained with visual materials. It was explained how to care for the episiotomy area to heal more rapid and healthier.
  * Information was given on how to change their menstrual pads.
  * Information was provided on what to look for when using underwear
  * What to watch out while taking a bath:
  * What to pay attention to in your stitch area
  Arms: training + written and illustrated training brochure

SUMMARY:
The World Health Organization (WHO) and professional societies recommend restricted episiotomy instead of routine episiotomy. However, since the 1990s, there has been evidence of the risks of the procedure, and although routine use has no benefit, it is still widely used. In this study, investigators aimed to determine the effect of episiotomy on the wound healing process and pain perception by providing episiotomy wound healing and genital hygiene training with training material created to raise awareness about wound care after episiotomy and to eliminate factors that delay the healing of episiotomy wound.

DETAILED DESCRIPTION:
This study aimed to determine the effect of episiotomy wound care and genital hygiene training on episiotomy wound healing and pain perception.

Methods: In this study, investigators used a randomized controlled trial approach.

It was carried out in the postpartum service of the medical faculty hospital. 128 participants who underlap vaginal postpartum episiotomy were randomly assigned to the experimental and control group. The women who gave birth in the experimental group were given episiotomy wound care and genital hygiene training. The routine postpartum care was given to the participants who gave birth in the control group. The data were collected using the personal information form, the episiotomy area evaluation scale (REEDA score), and the Visual Analog Scale (VAS).

.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* primiparous
* givingbirth vaginally on due date (37-42 gestational weeks)
* who have a healthy newborn,
* who have a mediolateral episiotomy,
* who do not have communication problems
* who can understand and speak Turkish were included in the research.

Exclusion Criteria:

* Givingbirth by cesarean section
* Having third and fourth-degree perineal tears,
* Having a history of diseases that prevent wound healing,
* Using certain drugs (eg, glucocorticoids, anticoagulants, chemotherapy, immunosuppressant, and radiotherapy),
* Having chronic systemic diseases (heart, kidney and lung diseases, coagulation disorder, immunodeficiency, connective tissue disorders, and diabetes),
* Having history of genital warts, symptomatic vaginitis,
* Having history of perineal reconstructive surgery, any postpartum complication (hemorrhage, puerperal infection, mastitis, thromboembolic disease or postpartum psychiatric disorder)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — 18 years of age and older primiparous women, who have given vaginally on the due date (37-42 gestational weeks) and have a mediolateral episiotomy
Enrollment: 128 (Actual)
Dates: Start 2022-03-03 (Actual); Primary Completion 2022-04-20 (Actual); Study Completion 2022-04-22 (Actual)

PRIMARY OUTCOMES:
Personal information form before intervention | postpartum 1sth day (after birth first 24 hours)
  Assessed using personal information. This instrument contains questions on women's sociodemographic and postpartum.
Episiotomy Area Evaluation before intervention | postpartum 1sth day (after birth first 24 hours)
  Assessed using the Episiotomy Area Evaluation Scale (REEDA SCORE) before intervention. This scale covers five factors indicating perineal wound healing: (1) Redness, (2) Edema, (3) Ecchymosis, (4) Discharge, and (5) Approximation. A total REEDA score is obtained by evaluating each category of these five recovery factors. The scale is evaluated by giving 0, 1, 2, and 3 points to each evaluation. The lowest score is 0 and the highest score is 15.
Episiotomy pain Evaluation before intervention | postpartum 1sth day (after birth first 24 hours)
  The Visual Analogue Scale (VAS) scale, which would be applied to evaluate episiotomy pain in the postpartum period, was used to convert some values that cannot be measured numerically, and two-end definitions of the parameter to be evaluated are written at both ends of a 100 mm line. The participant was asked to indicate where his or her condition is suitable on this line by drawing a line or by placing a dot or pointing. "No pain" is written on one end and "very severe pain" on the opposite end; the participant was asked to mark the pain condition on this line.was used to convert some values that could not be measured numerically, and two-end definitions of the parameter to be evaluated are written at both ends of a 100 mm line.

SECONDARY OUTCOMES:
Episiotomy Area Evaluation after intervention | postpartum 5th day
  Assessed using the Episiotomy Area Evaluation Scale (REEDA SCORE) before intervention. This scale covers five factors indicating perineal wound healing: (1) Redness, (2) Edema, (3) Ecchymosis, (4) Discharge, and (5) Approximation. A total REEDA score is obtained by evaluating each category of these five recovery factors. The scale is evaluated by giving 0, 1, 2, and 3 points to each evaluation. The lowest score is 0 and the highest score is 15.
Episiotomy pain Evaluation after intervention | postpartum 5th day
  The Visual Analogue Scale (VAS) scale, which would be applied to evaluate episiotomy pain in the postpartum period, was used to convert some values that cannot be measured numerically, and two-end definitions of the parameter to be evaluated are written at both ends of a 100 mm line. The participant was asked to indicate where his or her condition is suitable on this line by drawing a line or by placing a dot or pointing. "No pain" is written on one end and "very severe pain" on the opposite end; the participant was asked to mark the pain condition on this line.was used to convert some values that could not be measured numerically, and two-end definitions of the parameter to be evaluated are written at both ends of a 100 mm line.
Episiotomy Area Evaluation after intervention | Postpartum 15th day
  Assessed using the Episiotomy Area Evaluation Scale (REEDA SCORE) before intervention. This scale covers five factors indicating perineal wound healing: (1) Redness, (2) Edema, (3) Ecchymosis, (4) Discharge, and (5) Approximation. A total REEDA score is obtained by evaluating each category of these five recovery factors. The scale is evaluated by giving 0, 1, 2, and 3 points to each evaluation. The lowest score is 0 and the highest score is 15.
Episiotomy pain Evaluation after intervention | Postpartum 15th day
  The Visual Analogue Scale (VAS) scale, which would be applied to evaluate episiotomy pain in the postpartum period, was used to convert some values that cannot be measured numerically, and two-end definitions of the parameter to be evaluated are written at both ends of a 100 mm line. The participant was asked to indicate where his or her condition is suitable on this line by drawing a line or by placing a dot or pointing. "No pain" is written on one end and "very severe pain" on the opposite end; the participant was asked to mark the pain condition on this line.was used to convert some values that could not be measured numerically, and two-end definitions of the parameter to be evaluated are written at both ends of a 100 mm line.

CONTACTS AND LOCATIONS:
Overall Officials: Gonca Buran, PhD, Principal Investigator — Uludag Üniversity; Seyhan Çankaya, Ass. Prof, Study Chair — Selcuk University
Locations (1):
- Gonca Buran, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The data sets generated during and/or analyzed during the current study are available from the corresponding author on reasonable request.
Supporting Information: CSR
Time Frame: 6 months after publication
Access Criteria: relevance to the topic of the study and approval of all co-authors within 1 month of receiving the request.